CLINICAL TRIAL: NCT00624494
Title: Single Transpulmonary Thermodilution and Continuous Monitoring of Central Venous Oxygen Saturation During Off-pump Coronary Surgery
Acronym: OPCAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Mikhail Y. Kirov, Prof. M.Y. Kirov, MD, PhD, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4347.07.2006; Grant 4347.07.2006 (Other: HelseNord)
Record Dates: First submitted 2008-02-13; First posted 2008-02-27 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Hemodynamic Monitoring; Goal Directed Therapy
Keywords: venous oxygen saturation; transpulmonary thermodilution
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional monitoring (Active Comparator): hemodynamic monitoring - conventional monitoring
  Interventions: Device: Conventional monitoring
- Advanced monitoring (Active Comparator): hemodynamic monitoring - advanced monitoring
  Interventions: Device: Advanced monitoring

INTERVENTIONS:
Device: Conventional monitoring — In the CM group, therapy was guided by central venous pressure, mean arterial pressure (MAP) and heart rate (HR)
  Other Names: Non actual
  Arms: Conventional monitoring
Device: Advanced monitoring — In the AM group by the intrathoracic blood volume index, MAP, HR, central venous oxygen saturation (ScvO2) and cardiac index (CI). The measurements were performed before and during surgery, and at 2, 4 and 6 hrs post-operatively.
  Other Names: PiCCO-CeVOX
  Arms: Advanced monitoring

SUMMARY:
The aim of the present study was to evaluate the usefulness of an algorithm based on hemodynamic parameters obtained by single transpulmonary thermodilution (STD) combined with continuous monitoring of central venous oxygen saturation (ScvO2) for perioperative management of patients undergoing OPCAB.

DETAILED DESCRIPTION:
At the present time, there is an increasing tendency to perform off-pump coronary artery bypass grafting (OPCAB). However, OPCAB poses a variety of challenges from the point of view of the anesthesiologist and the intensivist. The aim of the present study was to evaluate the usefulness of an algorithm based on hemodynamic parameters obtained by single transpulmonary thermodilution (STD) combined with continuous monitoring of central venous oxygen saturation (ScvO2) for perioperative management of patients undergoing OPCAB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease, ranked ASA II-III and scheduled for elective OPCAB

Exclusion Criteria:

* Age < 18 years
* Severe valve dysfunction or peripheral vascular disease
* Simultaneous interventions (carotid endarterectomy, aneurysm repair, etc.)
* Transfer to CPB during surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | one month
  Length of the hospital stays, Days

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y Kirov, Study Director — Northern SMU
Locations (1):
- Dep. of Anesthesiology, Northern SMU, Arkhangelsk, Russia

REFERENCES:
- [Result] Smetkin AA, Kirov MY, Kuzkov VV, Lenkin AI, Eremeev AV, Slastilin VY, Borodin VV, Bjertnaes LJ. Single transpulmonary thermodilution and continuous monitoring of central venous oxygen saturation during off-pump coronary surgery. Acta Anaesthesiol Scand. 2009 Apr;53(4):505-14. doi: 10.1111/j.1399-6576.2008.01855.x. Epub 2009 Jan 15. PMID 19183113